CLINICAL TRIAL: NCT03386136
Title: Therapeutic Oxygen for Gastrointestinal Atony (TOGA): Pilot Trial - Management of Acute Colonic Pseudo-Obstruction With Oxygen Supplementation
Brief Title: Therapeutic Oxygen for Gastrointestinal Atony (TOGA)
Acronym: TOGA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB201701709
Record Dates: First submitted 2017-11-28; First posted 2017-12-29 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Ileus; Ogilvie Syndrome; Small Bowel Obstruction
Keywords: bowel ischemia; bowel perforation
MeSH Terms: conditions — Ileus; Colonic Pseudo-Obstruction; Intestinal Perforation | interventions — Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hospitalized Ileus or Pseudo-Obstruction Patient (Experimental): Hospitalized inpatient diagnosed with ileus, bowel obstruction or colonic pseudo-obstruction [clinician interpretation or small bowel diameter ≥3.5 cm, cecal diameter ≥ 9 cm, sigmoid colon diameter ≥ 6 cm] provided with 100% oxygen via non-rebreather face mask, for 6 hours
  Interventions: Drug: 100% Oxygen

INTERVENTIONS:
Drug: 100% Oxygen — To provide hospitalized ileus or pseudo-obstruction patient with 100% oxygen via non-rebreather face mask, for 6 hours

SUMMARY:
This study is a non invasive study to see if 100% oxygen therapy will help to resolve an intestinal obstruction.

DETAILED DESCRIPTION:
TOGA involves the provision of a 6- hour treatment with 100% oxygen via non breather mask to hospitalized patients with ileus, small bowel obstruction and/or colonic pseudo-obstruction will be a useful supplemental therapy, decreasing the diameter of the intestinal lumen and enhancing resolution of ileus/pseudo-obstruction

ELIGIBILITY:
Inclusion Criteria:

* patient or health proxy has been adequately informed of risks and benefits and agrees to his/her participation in the study.
* patient is a hospitalized inpatient diagnosed with ileus, bowel obstruction or colonic pseudo-obstruction [clinician interpretation or small bowel diameter ≥3.5 cm, cecal diameter ≥ 9 cm, sigmoid colon diameter ≥ 6 cm].
* patient is clinically and hemodynamically stable
* patient does not require supplemental oxygen greater than 2 liters per minute via nasal cannula
* patient does not have any respiratory contraindications to 100% oxygen
* failure to respond to non-surgical/non-endoscopic therapy for at least 24 hours, therapy at discretion of treating physician [to eliminate patients with trivial ileus not requiring advanced intervention]

Exclusion Criteria:

* patient is not expected to survive in the short term.
* patient is a pregnant or lactating woman.
* patient presents with severe or unstable psychiatric disorders.
* patient is participating in concomitant research studies that would interfere with this study.
* patient is an alcohol or drug abuser.
* respirator support required.
* unable to tolerate 100% oxygen for respiratory reasons or any other reasons.
* perforation of the viscus.
* inability to obtain informed consent.
* hypoxemia, as in room air oxygen saturation less than 90%.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2019-10-17 (Actual); Study Completion 2019-10-17 (Actual)

PRIMARY OUTCOMES:
Changes in Diameter of Colon | 6 - 24 hours
  X-ray of kidney, ureter and bladder (KUB) to determine maximal cecal diameter, maximal mid-transverse colon diameter, maximal mid-sigmoid colon diameter.
Changes in Diameter of the Small Bowel | 6 - 24 hours
  X-ray of kidney, ureter and bladder (KUB) to determine maximal cecal diameter, maximal mid-transverse colon diameter, maximal mid-sigmoid colon diameter.

SECONDARY OUTCOMES:
Demonstrates No Resolution of Ileus | 24 - 30 hours after initial TOGA
  A second treatment with TOGA will be offered.
Worsening of Ileus | 24 - 30 hours after initial TOGA
  Worsening of ileus after initial treatment but not requiring surgical or endoscopic intervention, will be offered a second treatment of TOGA.
Need for endoscopic or surgical intervention | 24 - 30 hours after initial TOGA
  Worsening of ileus after initial treatment, requiring surgical or endoscopic intervention
Length of Hospital Stay | up to 100 weeks
  Length of stay, measured at the end of hospitalization
Patient Complaints | Up to 48 hours
  Recording of patient perception/tolerance [daily] of TOGA.
Patient Pain Measurement | Up to 48 hours
  Patient pain measurement determined subjectively through a visual analogue scale (VAS) scale of 0 (no pain) to 10 (worst pain imaginable) taken before and after TOGA treatment.
Medication Measurement | 24 hours before through 24 hours after TOGA
  Documenting medication requirements for patients exposed to TOGA.(past 24 hours on a scale of 0 (no pain) to 10 (worst pain imaginable)

CONTACTS AND LOCATIONS:
Overall Officials: Brian C. Weiner, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Derived] Weiner B, Forsmark C, Khular V, Bauman A, Sutchu S, Banerjee D, Westerveld D, Zhang W, Jacobson M, Grajo J. TOGA Therapeutic Oxygen for Gastrointestinal Atony. Gastro Hep Adv. 2024 Jan 3;3(3):402-409. doi: 10.1016/j.gastha.2023.12.013. eCollection 2024. PMID 39131150